CLINICAL TRIAL: NCT05024734
Title: Guidance of Adjuvant Instillation in Intermediate Risk Non-muscle Invasive Bladder Cancer by Drug Screens in Patient Derived Organoids. A Single Center, Open-label, Phase II Trial With a Feasibility Endpoint. (GAIN-INST-TRIAL)
Brief Title: Guiding Instillation in Non Muscle-invasive Bladder Cancer Based on Drug Screens in Patient Derived Organoids
Acronym: GAIN INST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roland Seiler-Blarer (Other)
Collaborators: University of Bern (Other); Hospital Centre Biel/Bienne (Other)
Responsible Party: Sponsor-Investigator, Roland Seiler-Blarer, Chairman, Hospital Centre Biel/Bienne
Organization: Hospital Centre Biel/Bienne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZB-URO-21-001
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer; Non-muscle Invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Epirubicin; Mitomycin; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Epirubicin (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Epirubicin.
  If no significant drug selection can be performed in-vitro, Epirubicin will be the default for instillation.
  Interventions: Drug: Epirubicin
- Mitomycin (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Mitomycin.
  Interventions: Drug: Mitomycin
- Gemcitabine (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Gemcitabine.
  Interventions: Drug: Gemcitabine
- Docetaxel (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Docetaxel.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Epirubicin — In PDOs from patients that show highest response to Epirubicin, this drug will be instilled intravesically once weekly for 6 times.
  Epirubicin is also the default drug, in case of failure of drug prediction in the in-vitro drug screen in PDO.
  Epirubicin will be used as a concentrate for injection/instillation 2 mg/ml in total 50mg per vial. Prior to use, the concentrate for injection is diluted with 25ml of 0.9% saline solution to obtain the final Solution with 1mg/ml of Epirubicin.
  Arms: Epirubicin
Drug: Mitomycin — In PDOs from patients that show highest response to Mitomycin, this drug will be instilled intravesically once weekly for 6 times.
  Mitomycin C will be used as 20mg dry powder. Prior to use, the powder will be dissolved in 50ml of 0.9% saline solution according to the manufacturer instructions
  Arms: Mitomycin
Drug: Gemcitabine — In PDOs from patients that show highest response to Gemcitabine, this drug will be instilled intravesically once weekly for 6 times.
  Gemcitabine will be used as 2000 mg/50ml. For intravesical application, 1000mg of gemcitabine (corresponding to 25ml) will be diluted in 25ml 0.9% saline solution, to obtain the gemcitabine concentration of 1000mg/50ml used for instillation.
  Arms: Gemcitabine
Drug: Docetaxel — In PDOs from patients that show highest response to Docetaxel, this drug will be instilled intravesically once weekly for 6 times.
  Docetaxel will be used as 140mg/7ml solution. For intravesical application, 48.825ml of saline will be added to 1.875ml Docetaxel solution (according 37.5mg of Docetaxel). The concentration of this solution is 0.74mg/ml by a total volume of the instillation solution of 50,7.
  Arms: Docetaxel

SUMMARY:
From patients with intermediate risk non-muscle invasive bladder cancer tumor (NMIBC) specimens will be harvested during transurethral resection. Fresh specimens will be cultured as patient derived organoids (PDO). After approx. 10 days, PDO are exposed to different drugs that are used as intravesical instillation agents in these patients (epirubicin, mitomycin, gemcitabine, docetaxel). After 2 days of exposure, PDO viability will be measured. The drug with the highest antitumor effect on PDO will be applied as weekly intravesical instillations 6 times. Thereafter, patients are followed according to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent Form
* ECOG performance status of 0 or 1
* Histologically confirmed intermediate risk non muscle-invasive urothelial carcinoma of the bladder (pTa low grade) Patients
* Representative fresh tumor specimen for PDO generation and drug screen

Exclusion Criteria:

* Known previous high grade and/or high risk non muscle-invasive bladder cancer
* Previous Intravesical biological/immuno (BCG) therapy
* Pregnancy or nursing
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol
* Severe infection within 4 weeks prior to cycle 1, day 1
* Contraindication for frequent catheterization
* Voiding dysfunction
* Pregnancy or nursing
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 6 months after the last treatment.
* Male subject who is unwilling to use acceptable method of effective contraception during IP treatment and through 6 months after the last dose of IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with successful drug selection | 24 months
  Proportion of patients for which a specific selection of chemotherapeutic agent for intravesical instillation can be determined by using drug screens in PDOs.

SECONDARY OUTCOMES:
Proportion of patients for whom patient-derived organoids (PDOs) can be successfully generated (regardless of subsequent drug screen) | 24 months
  Proportion of patients for whom patient-derived organoids (PDOs) can be successfully generated (regardless of subsequent drug screen)
Rate of recurrence in the study population | 24 months
  Rate of recurrence in the study population
Recurrence free survival 24 months after TURBT | 24 months
  Proportion of patients that show recurrence 24 months after TURBT
Progression free survival 24 months after TURBT | 24 months
  Proportion of patients that show progression 24 months after TURBT
General quality of Life | 24 months
  Description of the general quality of life based on the questionnaire EORTC-QLQ-C30
Quality of Life related to the bladder cancer | 24 months
  Description of the Quality of Life related to the bladder cancer based on the specific NMIBC24 module
Safety profile of instillations | 24 months
  Description of the side effects related to the chemotherapeutic intravesical instillations occuring during the treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Seiler-Blarer, MD, Study Chair — Department of Urology
Locations (1):
- Spitalzentrum Biel/Bienne, Biel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Seiler R, Egger M, De Menna M, Wehrli S, Minoli M, Radic M, Lyatoshinsky P, Hosli R, Blarer J, Abt D, Kruithof-de Julio M. Guidance of adjuvant instillation in intermediate-risk non-muscle invasive bladder cancer by drug screens in patient derived organoids: a single center, open-label, phase II trial. BMC Urol. 2023 May 11;23(1):89. doi: 10.1186/s12894-023-01262-1. PMID 37170307